CLINICAL TRIAL: NCT07006493
Title: A Prospective, Multicenter, Randomized, Parallel-Controlled Superiority Study Evaluating the Efficacy and Safety of a Transcatheter Intramyocardial Septal Radiofrequency Ablation System in Patients With Obstructive Hypertrophic Cardiomyopathy
Brief Title: REFINE-HCM: Intramyocardial Septal Radiofrequency Ablation for Obstructive Hypertrophic Cardiomyopathy
Acronym: REFINE-HCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SuZhou Sinus Medical Technologies Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRCT-001
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Cardiomyopathy, Obstructive
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors are blinded to group assignment until completion of the 6-month primary endpoint assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Septal RF Ablation Group (Experimental): Participants in this group will receive a transcatheter intramyocardial septal radiofrequency ablation under intracardiac echocardiography (ICE) guidance using the investigational device system. Standardized pharmacological therapy will be continued throughout the study period.
  Interventions: Device: Transcatheter Intramyocardial Septal Radiofrequency Ablation System
- Sham Procedure (No RF Ablation) (Sham Comparator): Participants in this group will undergo a sham procedure under ICE guidance. The catheter will be inserted but no ablation will be performed. Participants will continue standardized pharmacological therapy throughout the study period. After completion of the 6-month follow-up, participants in this arm may voluntarily choose to receive the investigational treatment.
  Interventions: Device: Transcatheter Intramyocardial Septal Radiofrequency Ablation System

INTERVENTIONS:
Device: Transcatheter Intramyocardial Septal Radiofrequency Ablation System — The device system includes a single-use RF ablation catheter, sheath, RF generator, and irrigation pump. Ablation is guided by intracardiac echocardiography (ICE).

SUMMARY:
This is a prospective, multicenter, randomized, parallel-controlled, superiority clinical trial designed to evaluate the efficacy and safety of a transcatheter intramyocardial septal radiofrequency ablation system for the treatment of patients with obstructive hypertrophic cardiomyopathy (oHCM). Eligible participants will be randomized in a 2:1 ratio to receive either active ablation under intracardiac echocardiographic guidance or a sham procedure. All participants will continue to receive standard-of-care medical therapy during the study period. The primary endpoint is the treatment effectiveness rate at 6 months, defined as a ≥50% reduction in LVOT gradient from baseline or a resting LVOT gradient <30 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, regardless of sex
* Diagnosed with obstructive hypertrophic cardiomyopathy (oHCM)
* Presence of significant symptoms (e.g., dyspnea, chest pain, fatigue, palpitations, syncope)
* NYHA class II or higher with LVOTG ≥50 mmHg at rest or provoked (assessed by echocardiography)
* Septal thickness ≥15 mm
* Unsuitable for surgical myectomy or refusal of surgery
* Provided informed consent and agree to complete follow-up

Exclusion Criteria:

* Asymptomatic or non-obstructive HCM
* Septal thickness ≥30 mm
* Mitral valve anatomy not suitable for ablation as judged by investigator
* High risk of sudden cardiac death (SCD) requiring ICD implantation
* Complete right bundle branch block at screening
* Infective endocarditis, myocarditis, atrial myxoma, or intracardiac thrombus
* Contraindication to transseptal access (e.g., septal patch)
* Mechanical valves or history of aortic valve replacement
* Severe heart failure with persistent symptoms and LVEF <40%
* Major cardiac events within 6 months (e.g., cardiac arrest, MI, heart failure hospitalization)
* Significant structural heart disease requiring surgery
* Prior septal reduction therapy or pacemaker implantation
* Constrictive pericarditis or significant congenital heart disease
* Bleeding disorders or contraindication to antithrombotic therapy
* Liver dysfunction (ALT/AST >3× ULN)
* Renal insufficiency (creatinine >2.0 mg/dL or on dialysis)
* Pregnant, breastfeeding, or planning pregnancy within 6 months post-op
* Life expectancy <12 months
* Participation in other investigational studies within 30 days or 5 half-lives
* Investigator determines poor compliance or unsuitability
* Contraindications to cardiac MRI (e.g., ICD, allergy to contrast, claustrophobia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Effectiveness Rate at 6 Months | 6 months post-procedure
  Defined as either (1) a ≥50% reduction in resting LVOT gradient from baseline, or (2) resting LVOT gradient <30 mmHg.

SECONDARY OUTCOMES:
Change in Resting LVOT Gradient | Baseline, 6 months, 12 months
  Measured by echocardiography at baseline, 6 months, and 12 months
Change in NYHA Functional Class | Baseline, 6 months, 12 months
  Proportion of patients with improvement of ≥1 NYHA class
Change in 6-Minute Walk Distance | Baseline, 6 months, 12 months
  Distance walked in 6 minutes, compared to baseline
Change in 12-Item Short Form Health Survey (SF-12) Score | Baseline, 6 months, 12 months
  The SF-12 Health Survey includes two components: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores range from 0 to 100, with higher scores indicating better health status.
Device Success Rate | Day of procedure
  Defined as successful completion of RF ablation per protocol
Incidence of Adverse Events | Through 12 months
  All adverse events related to device or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Changshen Ma, Doctor, Principal Investigator — Capital Medical University Affiliated Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Capital Medical University Affiliated Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Sir Run Run Shaw hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) for this study.